CLINICAL TRIAL: NCT01054235
Title: Evaluation of Prenatal Care Program in Rural China
Brief Title: Prenatal Care Program in Dingyuan County
Acronym: EPCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Shanghai Medical University, School of Public Health, China (Unknown)
Responsible Party: Elina Hemminki, National Institute for Health and Welfare, Finland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 199901118
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Prenatal Care
Keywords: prenatal care; community-based randomized controlled trial; perinatal mortality; China
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- experimental (Experimental): The intervention consisted of 1) training township midwives, 2) informing women and men in the community of the importance of prenatal care, 3) providing intervention township hospitals with basic medical instruments used in prenatal care (i.e. blood pressure monitors, weighing scales for mothers and newborns, stethoscopes). For control ,none of the intervention will be given.
  Interventions: Behavioral: training

INTERVENTIONS:
Behavioral: training — The intervention consisted of 1) training township midwives, 2) informing women and men in the community of the importance of prenatal care, 3) providing intervention township hospitals with basic medical instruments used in prenatal care (i.e. blood pressure monitors, weighing scales for mothers and newborns, stethoscopes).

SUMMARY:
The general objective of this study is to evaluate prenatal care in the specific context of rural China. It also aims to define the optimal content of prenatal care for the context of rural China, to evaluate the effect of such prenatal care on infant and maternal outcomes, using a community based, well designed controlled trial in rural counties. Finally, it aims to describe the process of conducting a controlled study using community resources.

DETAILED DESCRIPTION:
The study was conducted in a rural county of 900,000 people in Anhui province, in eastern China. The total area of the county is almost 3,000 square kilometres. The majority of the population of the county is engaged in farming. In terms of national GDP rankings, the study county is typical of less developed rural areas in China. Twenty townships (10 interventions and 10 control) out of a total of 55 were selected - on the basis of having sufficient health facilities and staff - for a controlled trial on the introduction of systematic prenatal care in the area.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman in program area (in 20 townships) from August 2000 to March 2003

Exclusion Criteria:

* outsiders of program area

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Actual)
Dates: Start 2000-08; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
perinatal mortality | Jan 1999-Dec 2003

SECONDARY OUTCOMES:
timing and frequency of prenatal care and hospital delivery rate | Jan 1999-Dec 2003

CONTACTS AND LOCATIONS:
Overall Officials: Elina Hemminki, Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- County Health Bureau, Ding Yuan County, Chuzhou, Anhui, China

REFERENCES:
- [Result] Hemminki E, Wu Z, Cao G, Viisainen K. Illegal births and legal abortions--the case of China. Reprod Health. 2005 Aug 11;2:5. doi: 10.1186/1742-4755-2-5. PMID 16095526
- [Result] Wu Z, Viisainen K, Hemminki E. Determinants of high sex ratio among newborns: a cohort study from rural Anhui province, China. Reprod Health Matters. 2006 May;14(27):172-80. doi: 10.1016/S0968-8080(06)27222-7. PMID 16713892
- [Result] Wu Z, Viisainen K, Li X, Hemminki E. Maternal care in rural China: a case study from Anhui province. BMC Health Serv Res. 2008 Mar 10;8:55. doi: 10.1186/1472-6963-8-55. PMID 18331626
- [Result] Wu Z, Viisainen K, Wang Y, Hemminki E. Perinatal mortality in rural China: retrospective cohort study. BMJ. 2003 Dec 6;327(7427):1319. doi: 10.1136/bmj.327.7427.1319. PMID 14656839
- [Derived] Wu Z, Viisainen K, Wang Y, Hemminki E. Evaluation of a community-based randomized controlled prenatal care trial in rural China. BMC Health Serv Res. 2011 May 4;11:92. doi: 10.1186/1472-6963-11-92. PMID 21542939